CLINICAL TRIAL: NCT07393061
Title: Partial Wrist Denervation in Comminuted Articular Distal Radius Fractures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Momen Moustafa, professor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: denervation in fracture radius
Record Dates: First submitted 2026-01-22; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Parial Denervation; Fracture Disatl Radius
Keywords: parital denervation; comminuted distal radius fractures; chronic wrist pain

STUDY DESIGN:
Intervention Model Description: observational
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- parital wrist denervation (Other): Partial Wrist Denervation in Comminuted articular Distal Radius Fractures
  Interventions: Procedure: Partial Wrist Denervation in Comminuted articular Distal Radius Fractures

INTERVENTIONS:
Procedure: Partial Wrist Denervation in Comminuted articular Distal Radius Fractures — Partial Wrist Denervation in Comminuted articular Distal Radius Fractures through sme approach of the surgery

SUMMARY:
the aim of Partial Wrist Denervation in Comminuted articular Distal Radius Fractures is to decrease incidence of chronic wrist pain follwing this type of fracture

DETAILED DESCRIPTION:
Distal radius fractures represent the most common fractures in adults showing an overall prevalence of 17.5 % with respect to all fractures. partial wrist denervation is an adjunctive procedure performed during initial fracture fixation to mitigate chronic pain by interrupting sensory innervation to the wrist joint. It targets the anterior interosseous nerve (AIN) and posterior interosseous nerve (PIN), which convey nociceptive signals from the radiocarpal and midcarpal joints.

Comminuted intra-articular distal radius fractures (AO/OTA Type C2/C3) often lead to post-traumatic arthritis due to articular incongruity and capsular damage. Denervation at the index procedure may reduce central sensitization and chronic pain by resecting afferent pain fibers, potentially improving postoperative rehabilitation and functional outcomes.

Acute comminuted intra-articular distal radius fractures (AO/OTA C2/C3) with high risk of post-traumatic arthritis (e.g., articular step-off >2 mm, severe fragmentation).

* Active individuals seeking motion preservation, those with high functional demands (e.g., athletes, laborers), or patients preferring a less invasive option than salvage procedures.
* Adjunct to primary fixation: Performed concurrently with volar locking plate (VLP) or dorsal plating.

ELIGIBILITY:
Inclusion Criteria:• Age from 18

* Fracture Pattern: Acute, comminuted intra-articular distal radius fractures (AO/OTA Type C2 or C3).
* Surgical Context: Procedure performed as a primary adjunct during initial open reduction and internal fixation (ORIF).

Exclusion Criteria:Active local infection over the surgical site.

* Compromised soft tissue envelope that precludes safe dissection.
* Vascular injury or compromise requiring repair.
* Pre-existing neurological deficit (e.g., complex regional pain syndrome, major peripheral nerve injury).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The end results PAIN will be assessed according to mayo clinc wrist score | 2 weeks, 6 weeks, 3 months, 6 months..and 1 year
  mayo clinc wrist score its a clincal reported outcome measure designed to assess function and pain of the wrist follwing surgery the score is bassed on 100 points divided into four equally weighted categories the final score places the wrist into outcome category total score 90/100 is excellent while below 65 is poor

CONTACTS AND LOCATIONS:
Overall Officials: walyd ryad saleh, professor of orthopedics, Study Director — Assiut University
Locations (1):
- Assiut Universty, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
will wait till we see the result

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/citmatch/